CLINICAL TRIAL: NCT05048238
Title: Evaluation of Tofacitinib in Prevention of Photosensitivity in Cutaneous Lupus Erythematosus (ALE11)
Brief Title: Evaluation of Tofacitinib in Prevention of Photosensitivity in Lupus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ALE11
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cutaneous Lupus
Keywords: Systematic Lupus Erythematosus; Lupus; Systemic Lupus; Cutaneous Lupus; Tofacitinib; Ultraviolet
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tofacinitib (Experimental): 10 participants receiving 11 mg of Tofacitinib administered orally and daily, from Day 2 to Day 26
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — 10 participants with Cutaneous lupus erythematosus (CLE). Consenting individuals meeting all entry criteria will undergo 25 days of treatment with tofacitinib (11 mg orally (PO) daily) with evaluation of UVB-mediated cutaneous apoptosis
  Other Names: XELJANZ(R) XR

SUMMARY:
This is a single-arm, multi-site, proof-of-concept study that will evaluate the treatment of 10 participants with cutaneous lupus erythematosus (CLE) with Tofacitinib.

DETAILED DESCRIPTION:
Once consented, study participants meeting all entry criteria will undergo 25 days of treatment with tofacitinib (11 mg orally daily). Tofacitinib will be distributed to eligible participants at Visit 2 (Day 1) and the first dose will be taken on Day 2. The last dose is the morning of Visit 5 (Day 26).Ultraviolet B (UVB)-mediated cutaneous apoptosis and ancillary mechanistic studies will be evaluated in phototests, skin biopsies and blood samples collected before and after treatment.

This study will assess whether a 25-day regimen of tofacitinib impacts photosensitivity following UVB exposure in individuals with CLE.

ELIGIBILITY:
Inclusion Criteria:

1. Cutaneous lupus erythematosus based upon all of the following:

   1. a clinical diagnosis made by a rheumatologist or dermatologist of one of the following: acute cutaneous lupus erythematosus, subacute cutaneous lupus, or chronic cutaneous lupus erythematosus;
   2. active skin disease within 5 years prior to screening. Participants may have concomitant SLE.
2. SLEDAI-2K score ≤4 (clinical criteria only, excludes all laboratory criteria) for all participants regardless of whether they have concomitant SLE.
3. If taking oral corticosteroids, the dose must be ≤ 10 mg daily of prednisone (or equivalent), stable dose for at least 4 weeks, and not anticipated to change over the course of the study.
4. If taking oral anti-malarial medications, the dose(s) must be ≤ 100 mg daily for quinacrine or/and ≤ 400 mg daily for hydroxychloroquine, stable for at least 6 months, and not anticipated to change over the course of the study.
5. If taking oral or subcutaneous methotrexate, the dose must be ≤ 25 mg weekly, stable for at least 4 weeks, and not anticipated to change over the course of the study.
6. If taking oral leflunomide, the dose must be ≤ 20 mg daily, stable for at least 4 weeks, and not anticipated to change over the course of the study.
7. If taking oral mycophenolate mofetil (MMF) or mycophenolic acid, the dose must be equivalent to ≤ 3000 mg of MMF daily, stable for at least 4 weeks, and not anticipated to change over the course of the study.
8. Adults 18 to 65 years of age at screening.
9. All participants and/or their sexual partners who engage in sexual activity that could lead to pregnancy must be willing to use complete abstinence or an FDA-regulated form of contraception for the duration of the study and for at least one month after discontinuation of study drug to prevent pregnancy. Highly effective birth control methods include, but are not limited to, hormonal contraception, an intrauterine device, or surgical options. Periodic abstinence and withdrawal are not acceptable methods of birth control.

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
2. Current or recent history, within the last year, of uncontrolled clinically significant renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurologic disease or significant impairment that might negatively impact the participant's ability to participate or that may put a participant at increased risk.
3. Potential active nephritis and/or urinary tract infection at screening, defined as any one of the following determined at screening unless otherwise specified:

   1. >10 RBCs /hpf,
   2. >5 WBCs /hpf with either positive nitrites or greater than a trace leukocyte esterase,
   3. Signs or symptoms of a urinary tract infection,
   4. For individuals with no history of nephritis: Urine protein (mg/dL): creatinine (mg/dL) ratio (Pr/Cr)>0.5 at screening or a Pr/Cr level that has exceeded 1.0 in the prior 12 months,
   5. For individuals with a history of nephritis: A rise in Pr/Cr of >0.5 over the prior 3-6 months prior to screening.
4. History of severe gastrointestinal narrowing or strictures.
5. Medically confirmed history of diverticulitis or chronic, ulcerative lower gastrointestinal (GI) disease such as Crohn's disease, ulcerative colitis, or other symptomatic, lower GI conditions that might predispose a participant to perforations.
6. History of thrombosis, pulmonary embolism, or antiphospholipid syndrome.
7. History of any one of the following anti-phospholipid antibodies:

   1. Positive lupus anticoagulant test, or
   2. Anti-β2-glycoprotein I IgG ELISA titer ≥ 40 GPL, or
   3. Anti-cardiolipin IgG ELISA titer ≥ 40 GPL.
8. History of chronic pulmonary disease requiring supplemental oxygen including chronic obstructive pulmonary disease (COPD) requiring chronic treatment, interstitial lung disease (ILD) requiring immunosuppressive therapy, and asthma requiring chronic steroid (other than inhaled steroid) or biologic therapy.
9. History of moderate to severe atherosclerotic cardiovascular disease as evidenced by prior coronary artery bypass surgery, coronary artery stent placement, myocardial infarction, symptomatic carotid arterial disease, peripheral vascular disease, abdominal aortic aneurysm; or angina within the past 8 weeks prior to Visit 1 (Day 0).
10. History of keloid scarring.
11. History of any lymphoproliferative disorder or other malignancy with the exception of successfully treated or excised basal cell or squamous cell skin cancer or cervical cancer in situ.
12. Other autoimmune diseases likely to require immunosuppression.
13. Any of the following lab results at screening:

    1. Hemoglobin <9.5 g/dL
    2. White Blood Cell count <3.5 x 109/L
    3. Absolute Neutrophil count <1.2 x 109/L
    4. Platelet count <120 x 109/L
    5. Absolute Lymphocyte count <0.75 x 109/L
    6. Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 1.5 × the upper limit of normal (ULN)
    7. Total bilirubin > ULN
    8. Estimated glomerular filtration rate [GFR] <60mL/min/1.73 m2
    9. Triglycerides ≥ 300 mg/dL (fasting not required)
    10. Total Cholesterol ≥ 240 mg/dL (fasting not required).
14. Major surgery < 8 weeks prior to Visit 1 (Day 0).
15. Hospitalized for serious infection < 4 weeks prior to Visit 1 (Day 0).
16. Chronic infections other than chronic or intermittent uncomplicated urinary tract infections (including but not limited to tuberculosis, chronic pyelonephritis, osteomyelitis).
17. Presumed or documented COVID-19 infection within 30 days prior to Visit 1 (Day 0).
18. Recent (within one month prior to screening) close contact with a person who has active TB infection.
19. History of untreated active or latent TB infection.
20. History of incompletely treated active or latent TB infection unless at least one month of treatment has been completed prior to screening.
21. Positive Interferon-Gamma Release Assay (IGRA) or positive purified protein derivative tuberculin skin test (PPD) (> 5mm induration) at screening.
22. An indeterminate IGRA at screening unless followed by a subsequent negative IGRA or negative PPD.
23. History of human immunodeficiency virus (HIV).
24. A positive test for HIV antigen/antibody or nucleic acid test (NAT) at screening.
25. History of a hepatitis B infection.
26. A positive test for hepatitis B surface antigen or hepatitis B core antibody at screening.
27. History of a hepatitis C infection.
28. A positive test for hepatitis C antibody (regardless of whether hepatitis C RNA levels are undetectable) at screening.
29. History of recurrent (more than one episode) herpes zoster, one or more episodes of any of the following: herpes zoster ophthalmicus, or disseminated herpes zoster, or disseminated herpes simplex.
30. Current, recent (< 4 weeks prior to Visit 1 (Day 0)) or chronic use of antibiotic medication, except for suppression of chronic/recurrent urinary tract infection, which is allowed.
31. Simultaneous use of more than one of the following: leflunomide, methotrexate and MMF.
32. Any of the following active medications (oral or parenteral): cyclosporine, voclosporin, cyclophosphamide, tacrolimus, rituximab or other anti-CD20s, or any other investigational or marketed biologic with immunomodulatory properties within a year prior to Visit 1 (Day 0).
33. Any of the following medications (oral or parenteral): azathioprine or belimumab within 3 months prior to Visit 1 (Day 0).
34. Any prior treatment with cell-depleting therapies other than anti-CD20s including but not limited to CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 products.
35. Intravenous or intramuscular corticosteroids within 2 weeks prior to Visit 1 (Day 0).
36. Treatment with any investigational agent ≤ 4 weeks or ≤ 5 half-lives of the investigational drug prior to Visit 1 (Day 0), whichever is longer.
37. Treatment with more than one dose of ketoconazole within one week of screening.
38. Any prior treatment with chlorambucil, bone marrow transplantation, or total lymphoid irradiation.
39. Vaccinated or exposed by close contact, e.g., within a household, to a live/attenuated vaccine ≤ 6 weeks prior to Visit 1 (Day 0); or is expected to be vaccinated or to have household exposure to these vaccines during treatment or during the 6 weeks following discontinuation of study medication.
40. Received a non-live vaccine ≤ 2 weeks prior to initiation of study drug, or unwillingness of a participant to delay non-live vaccination until 1 month after completion of study therapy.
41. Pregnant or breastfeeding females.
42. History of alcohol or substance abuse, unless in full remission for greater than 6 months prior to first dose of study drug.
43. Past or current medical or psychiatric conditions or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Kahlenberg, M.D., Ph.D., Study Chair — University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology
Locations (2):
- United States (2):
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort [https://immport.niaid.nih.gov/ ], a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts, upon completion of the study.
Time Frame: After completion of the study
Access Criteria: Data will be sent to ImmPort, but not made available to the public, due to small sample size of study.
URL: http://www.immport.org/home

REFERENCES:
- See also: Autoimmunity Centers of Excellence (ACE) — http://www.autoimmunitycenters.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two study sites were activated in the United States, beginning in March 2022. A total of eight participants were screened from September 2022 to January 2024 at both sites. Of those screened seven participants enrolled in the study.
Groups:
- Tofacitinib: 25-day regimen of tofacitinib 11 mg daily
Period: Overall Study
Arm/Group | Tofacitinib
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Enrolled
Arm/Group | Tofacitinib
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (6.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Diagnosed with Systemic Lupus Erythematosus (SLE) [Count of Participants; unit: Participants] — Diagnosis of systemic lupus erythematosus (SLE) per ACR/EULAR criteria was confirmed at screening visit.
  Participants
    Yes | 3
    No | 4
Fitzpatrick Scale [Count of Participants; unit: Participants] — Participants were categorized by Fitzpatrick skin types - Type I being lightest and Type VI being darkest - at their screening visit.
  Participants
    Type I | 1
    Type II | 2
    Type III | 1
    Type IV | 2
    Type V | 1
    Type VI | 0
SLEDAI-2K Score (Clinical Criteria Only) [Mean (Standard Deviation); unit: SLEDAI-2K Score] — Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) is a validated, physician-based assessment tool used to measure the extent of lupus disease activity within the past 30 days. SLEDAI-2K total score is a weighted sum of the presence of 24 lupus disease symptoms and ranges from 0 to 105, with higher scores indicating more lupus disease activity present.For this assessment, only clinical criteria were considered; laboratory criteria were excluded.
  SLEDAI-2K Score | 0.9 (1.07)
CLASI Total Activity (CLASI-A) Score [Mean (Standard Deviation); unit: CLASI-A Score] — Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) is a validated, physician-based assessment tool used to measure cutaneous lupus severity. Severity is calculated based on disease activity (erythema and scale) and damage (dyspigmentation and scarring) for the cumulative areas of involved skin. CLASI activity score ranges from 0 to 70, with higher scores indicating increased disease severity.
  CLASI-A Score | 2.4 (3.87)
CLASI Total Damage (CLASI-D) Score [Mean (Standard Deviation); unit: CLASI-D Score] — CLASI is a validated, physician-based assessment tool used to measure cutaneous lupus severity. Damage is calculated based on dyspigmentation and scarring for the cumulative areas of involved skin. The CLASI damage score ranges from 0 to 56, with higher scores indicating worse damage to the skin due to lupus.
  CLASI-D Score | 2.9 (5.40)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of UVB-induced Apoptotic Epidermal Cells
Description: At Day 0 and Day 25, skin was exposed to 10-80 mJ/cm2 UVB irradiation. At Day 1 and Day 26, erythema levels were measured with a Chroma Meter at each dose site and in an unexposed section. Skin biopsies at Day 1 and Day 26 were taken at the unexposed site and at the minimal erythema dose (MED) at Day 1. The percentage of apoptotic epidermal cells were determined in each skin biopsy sample by TUNEL staining. The percentage of UVB-induced apoptotic cells is defined as the difference between the percentage of apoptotic epidermal cells in the UVB-exposed biopsy at the MED and percentage of apoptotic epidermal cells in the unexposed biopsy at the same visit. Change in percentage of UVB-induced apoptotic epidermal cells is calculated as the difference in the percentage of UVB-induced apoptotic cells at Day 26 and at Day 1.
Time Frame: Day 1 (pre-treatment) to Day 26
Population: The Per Protocol 1 (PP1) population includes all participants who received any amount of tofacitinib and who completed phototests and skin biopsies at both baseline (Visits 1 and 2) and post-treatment (Visits 4 and 5) time points. Only individuals who completed at least 21 days of IP dosing had the post-treatment phototest.
Measure: Mean (Standard Deviation); unit: percentage of epidermal cells
Arm/Group | Tofacitinib
Number analyzed (Participants) | 6
percentage of epidermal cells
  Day 1 | 20.06 (9.587)
  Day 26 | 3.03 (2.349)
  Change from Day 1 to Day 26 | -17.03 (8.355)

2. Primary Outcome: Change in Percentage of UVB-induced Apoptotic Epidermal Cells
Description: as for outcome 1
Time Frame: Day 1 (pre-treatment) to Day 26
Population: The Per Protocol 2 (PP2) population includes all PP1 participants with no protocol deviations that would impact photo sensitivity assessments.
Measure: Mean (Standard Deviation); unit: percentage of epidermal cells
Arm/Group | Tofacitinib
Number analyzed (Participants) | 3
percentage of epidermal cells
  Day 1 | 21.51 (12.334)
  Day 26 | 3.45 (2.976)
  Change from Day 1 to Day 26 | -18.06 (11.182)

3. Secondary Outcome: Change in Minimal Erythema Dose (MED) Due to UVB
Description: At Day 0 and Day 25, skin was exposed to 10-80 mJ/cm2 UVB irradiation. At Day 1 and Day 26, erythema levels were measured with a Chroma Meter at each dose site and in an unexposed section. The MED was defined as the dose that contained the lowest UVB exposure and the average redness reading that was at least 2.5 higher than the average redness reading in the unexposed skin. The possible values for MED ranged from 10 to 80 mJ/cm2.
Time Frame: Day 1 (pre-treatment) to Day 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 6
Participants
  +30 mJ/cm2 | 0
  +20 mJ/cm2 | 0
  +10 mJ/cm2 | 1
  Stayed the same | 3
  -10 mJ/cm2 | 0
  -20 mJ/cm2 | 1
  -30 mJ/cm2 | 1

4. Secondary Outcome: Change in UVB-induced Expression of Inflammatory Genes in Skin Based on Enumeration of RNA Transcripts.
Description: Skin biopsies at Day 1 and Day 26 were taken at the unexposed site and at the site corresponding to the next higher UVB dose than the Day 26 MED. RNA was isolated and expression values were analyzed by RNA sequencing. UVB-induced expression is defined as the difference in expression measured in the biopsy exposed at the Visit 2 (Day 1) 1x minimal erythema dose (MED) and that measured in the unexposed biopsy.
Time Frame: Day 1 (pre-treatment) to Day 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Count of RNA transcripts
Arm/Group | Tofacitinib
Number analyzed (Participants) | 6
Count of RNA transcripts
  TNF at Day 1 | -5.5 (10.13)
  TNF at Day 26 | -0.8 (5.85)
  TNF Change from Day 1 to Day 26 | 4.7 (6.50)
  IL1B at Day 1 | 38.5 (42.57)
  IL1B at Day 26 | 4.8 (20.82)
  IL1B Change from Day 1 to Day 26 | -33.7 (44.85)
  CXCL9 at Day 1 | 53.8 (63.35)
  CXCL9 at Day 26 | 133.7 (246.27)
  CXCL9 Change from Day 1 to Day 26 | 79.8 (289.29)
  IL6 at Day 1 | -0.7 (5.24)
  IL6 at Day 26 | 10.5 (25.74)
  IL6 Change from Day 1 to Day 26 | 11.2 (25.33)
  IFNB1 at Day 1 | 0.0 (0.00)
  IFNB1 at Day 26 | 0.00 (0.00)
  IFNB1 Change from Day 1 to Day 26 | 0.0 (0.00)
  IFI44 at Day 1 | 10.2 (54.62)
  IFI44 at Day 26 | 109.5 (137.50)
  IFI44 Change from Day 1 to Day 26 | 99.3 (107.08)

5. Secondary Outcome: Change in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score
Description: CLASI is a validated, physician-based assessment tool used to measure cutaneous lupus severity. Severity is calculated based on disease activity (erythema and scale) and damage (dyspigmentation and scarring) for the cumulative areas of involved skin. CLASI activity score ranges from 0 to 70, with higher scores indicating increased disease severity.
Time Frame: Day 0 (pre-treatment) to Day 25
Population: The Per Protocol 1 (PP1) population includes all participants who received any amount of tofacitinib and who completed phototests and skin biopsies at both baseline (Visits 1 and 2) and post-treatment (Visits 4 and 5) time points. Only individuals who complete at least 21 days of IP dosing had the post-treatment phototest.
Measure: Mean (Standard Deviation); unit: CLASI-A Score
Arm/Group | Tofacitinib
Number analyzed (Participants) | 6
CLASI-A Score
  Day 0 | 2.8 (4.07)
  Day 25 | 2.3 (3.27)
  Change from Day 0 to Day 25 | -0.5 (1.22)

6. Secondary Outcome: Change in CLASI Damage Score
Description: CLASI is a validated, physician-based assessment tool used to measure cutaneous lupus severity. Damage is calculated based on dyspigmentation and scarring for the cumulative areas of involved skin. The CLASI damage score ranges from 0 to 56, with higher scores indicating worse damage to the skin due to lupus.
Time Frame: Day 0 (pre-treatment) to Day 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CLASI-D Score
Arm/Group | Tofacitinib
Number analyzed (Participants) | 6
CLASI-D Score
  Day 0 | 3.3 (5.75)
  Day 25 | 2.8 (4.67)
  Change to Day 25 | -0.5 (1.22)

7. Secondary Outcome: Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Total Score
Description: Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) is a validated, physician-based assessment tool used to measure the extent of lupus disease activity within the past 30 days. SLEDAI-2K total score is a weighted sum of the presence of 24 lupus disease symptoms and ranges from 0 to 105, with higher scores indicating more lupus disease activity present.
Time Frame: Day 0 (pre-treatment) to Day 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SLEDAI-2K Score
Arm/Group | Tofacitinib
Number analyzed (Participants) | 6
SLEDAI-2K Score
  Day 0 | 1.3 (1.63)
  Day 25 | 1.7 (1.97)
  Change to Day 25 | 0.3 (0.82)

8. Secondary Outcome: Change in Severity Grade for Laboratory Tests From Grade 0
Description: The study sites graded the severity of laboratory results for the study participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) 5.0. The NCI-CTCAE manual provides a common language to describe levels of severity, to analyze and interpret data, and to articulate the clinical significance of adverse events. Select laboratory results are incorporated into relevant adverse event criteria.
Time Frame: Screening Visit through Day 40
Population: The Safety Sample (SS) population includes all participants who received any amount of tofacitinib.
Measure: Number; unit: participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 7
participants
  Alanine Aminotransferase: Increase by 1 grade | 1
  Alanine Aminotransferase: Increase by 2+ grades | 0
  Aspartate Aminotransferase: Increase by 1 grade | 1
  Aspartate Aminotransferase: Increase by 2+ grades | 0
  Total Cholesterol: Increase by 1 grade | 2
  Total Cholesterol: Increase by 2+ grades | 0

9. Secondary Outcome: Treatment-emergent Adverse Events by Severity
Description: The study sites graded the severity of AEs experienced by the study participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) 5.0. The NCI-CTCAE manual provides a common language to describe levels of severity, to analyze and interpret data, and to articulate the clinical significance of all AEs. A treatment-emergent AE is defined as an increase in grade from the last assessment prior to a participant starting treatment at Day 2, or from the last post-baseline value that doesn't meet grading criteria. AEs were classified by system organ class and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) version 25.1.
Time Frame: Day 2 to Day 40
Population: The Safety Sample (SS) population includes all participants who received any amount of tofacitinib.
Measure: Number; unit: Adverse Events
Arm/Group | Tofacitinib
Number analyzed (Participants) | 7
Adverse Events
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

10. Secondary Outcome: Treatment-emergent Adverse Events by Relationship to Tofacitinib
Description: The relationship, or attribution, of an adverse event to the study therapy regimen or study procedure(s) was initially determined by the site investigator and recorded on the appropriate AE/SAE eCRF as not related, possibly related or related. Final determination of attribution for safety reporting was determined by sponsor. An AE assessed as possibly related or related was classified as related to the study therapy or procedure. A treatment-emergent AE is defined as an increase in grade from the last assessment prior to a participant starting treatment at Day 2, or from the last post-baseline value that doesn't meet grading criteria. AEs were classified by system organ class and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) version 25.1.
Time Frame: Day 2 to Day 40
Population: The Safety Sample (SS) population includes all participants who received any amount of tofacitinib.
Measure: Number; unit: Adverse Events
Arm/Group | Tofacitinib
Number analyzed (Participants) | 7
Adverse Events
  Related to Tofacitinib | 0
  Not Related to Tofacitinib | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected in EDC from Day 2 until Day 40.
Description: Adverse events (AEs) of Grade 2 or higher and all Grade 1 or higher COVID-19 events were recorded in EDC. A treatment-emergent AE is defined as an increase in grade from the last assessment prior to a participant starting treatment at Day 2, or from the last post-baseline value that doesn't meet grading criteria. AEs were classified by system organ class and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) version 25.1.
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib (N=7)
Dental caries (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The protocol specified inferential statistics for the primary and some secondary endpoints. Given the small number of participants enrolled, no statistical testing was performed, and only descriptive statistics are presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05048238/Prot_SAP_003.pdf
  • Informed Consent Form (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05048238/ICF_002.pdf